CLINICAL TRIAL: NCT04468958
Title: A Phase 1, Randomized, Double-Blind, Placebo-Controlled, Single and Multiple Ascending Dose Study of SAB-185 in Healthy Subjects
Brief Title: Safety, Tolerability, and Pharmacokinetics of SAB-185 in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: SAb Biotherapeutics, Inc. (Industry)
Collaborators: Department of Health and Human Services (U.S. Federal Agency); JPEO, Chemical, Biological, Radiological, and Nuclear Defense (CBRND) Enabling Biotechnologies (EB) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SAB-185-101
Record Dates: First submitted 2020-07-08; First posted 2020-07-13 (Actual); Last update posted 2022-07-01 (Actual); Status verified 2022-06

CONDITIONS: COVID-19; SARS-CoV2
MeSH Terms: conditions — COVID-19 | interventions — SAB-185; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- 10mg/kg SAB-185 (Experimental): 10mg/kg SAB-185 in normal (0.9%) saline; concentration 4mg/mL (0.4%)
  Interventions: Biological: SAB-185
- 25mg/kg SAB-185 (Experimental): 25mg/kg SAB-185 in normal (0.9%) saline; concentration 20mg/mL (2%)
  Interventions: Biological: SAB-185
- 25mg/kg SAB-185 x 2 doses (Experimental): 25mg/kg SAB-185 in normal (0.9%) saline; concentration 20mg/mL (2%). Cohort 3 will receive a second 25mg/kg dose of SAB-185 7 days (+/-2) after the first treatment.
  Interventions: Biological: SAB-185
- 50mg/kg SAB-185 (Experimental): 50mg/kg SAB-185 in normal (0.9%) saline; concentration 20mg/mL (2%)
  Interventions: Biological: SAB-185
- Placebo (Placebo Comparator): Normal (0.9%) saline in approximately the same volume as each cohort in the experimental drug arm.
  Interventions: Other: Normal saline

INTERVENTIONS:
Biological: SAB-185 — SAB-185 is a purified human immunoglobulin G (hIgG) designed to specifically bind to Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-CoV-2) viruses. SAB-185 is purified from the plasma of immunized Tc bovines that were immunized initially (vaccinations 1 and 2) with a plasmid DNA (pDNA) vaccine that expresses wild-type SARS-CoV-2 spike protein, followed by additional immunizations (vaccinations 3 and beyond) with a recombinant spike protein from SARS-CoV-2 produced in insect cells. The purified hIgG is a sterile liquid formulated in 10 mM glutamic acid monosodium salt, 262 mM D-sorbitol, 0.05 mg/mL Tween 80, pH 5.5. The drug product will be administered intravenously and will be diluted in saline per the clinical protocol.
  Other Names: Anti-SARS-CoV-2 Human Immunoglobulin Intravenous (Tc bovine-derived)
  Arms: 10mg/kg SAB-185; 25mg/kg SAB-185; 25mg/kg SAB-185 x 2 doses; 50mg/kg SAB-185
Other: Normal saline — Normal (0.9%) saline in approximately the same volume as each cohort in the experimental drug arm.
  Arms: Placebo

SUMMARY:
Coronavirus disease 2019 (COVID-19) is an infectious disease caused by severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2). SAB Biotherapeutics has developed SAB-185, an Anti-SARS-CoV-2 Human Immunoglobulin Intravenous (transchromosomic [Tc] bovine-derived), as a potential therapeutic to treat COVID-19. This study will evaluate the safety, immunogenicity, and pharmacokinetics of SAB-185 in healthy participants.

DETAILED DESCRIPTION:
There were 4 treatment groups and 1 control group. Cohort 1 received 1 dose of SAB-185 at 10 mg/kg per dose. Cohort 2 received 1 dose of SAB-185 at 25 mg/kg, Cohort 3 received 2 doses of SAB-185 at 25 mg/kg each 7 days apart, and Cohort 4 received 1 dose of SAB-185 at 50 mg/kg per dose. All the doses were prepared at the site by the pharmacy staff or designee for delivery to the clinical staff for administration, per the site's SOPs.

ELIGIBILITY:
Inclusion Criteria:

Subjects must meet all of the following criteria for inclusion:

1. 18-60 years of age
2. Able to understand the study and comply with all study procedures
3. Agrees not to participate in any other trial of an investigational product during the study period
4. Willing and able to provide written informed consent prior to the start of any study related activities
5. In good health in the opinion of the site principal investigator as determined by vital signs, medical history, physical examination and clinical laboratory tests
6. If female, meets at least one of the following reproductive risk criteria

   * Post-menopausal for at least 12 months
   * Use of one or more of the following highly effective contraceptive methods for at least 90 days following the last dose of study product: combined estrogen and progestogen containing or progestogen-only hormonal contraception, intrauterine device (IUD), intrauterine hormone-releasing system, surgical bilateral tubal occlusion
   * Vasectomized sole sexual partner who has received medical assessment of the surgical success
7. Subjects agree to sexual abstinence (refraining from heterosexual intercourse for at least 90 days following the last dose of study product) if not using birth control or condoms for males.

Exclusion Criteria:

1. Female subjects with positive pregnancy test, breastfeeding, or planning to become pregnant/breastfeed during the study period.
2. Treatment or participation in another clinical trial of any other investigational agent within 30 days prior to enrollment.
3. Use of other drugs that, in the opinion of the investigator, could complicate analysis of SAB-185.
4. Subjects with the following risk factors:

   * Compromised immune system including confirmed diagnosis of current cancer under treatment, inherited deficiencies of the immune system, immune suppressing medication, or other conditions causing leukopenia or neutropenia
   * Known autoimmune condition requiring therapy more intensive than intermittent non-steroidal anti-inflammatories in the prior 6 months (for example: rheumatoid arthritis, lupus, inflammatory bowel disease)
   * Chronic respiratory disease including COPD, emphysema, cystic fibrosis, pulmonary hypertension, or other chronic condition that requires the routine use of supplemental oxygen
   * Chronic asthma requiring the use of oral steroids or hospitalization in the last six months
   * Renal failure or renal insufficiency requiring dialysis
   * Congestive heart failure or significant atherosclerotic disease (coronary artery disease or peripheral vascular disease)
   * Hypertension, diabetes, those currently vaping or smoking or with a history of chronic smoking, and those with BMI > 35 kg/m2
5. Receipt of pooled immunoglobulin or plasma in past 30 days
6. Any other underlying medical (cardiac, liver, renal, neurological, respiratory) or psychiatric condition that in the view of the investigator would preclude use of SAB-185
7. Known IgA deficiency or previous allergic reaction to intravenous immunoglobin (IVIG)/subcutaneous immunoglobin (SCIG)
8. Positive screening test for hepatitis B virus surface antigen, hepatitis C virus antibody, or HIV antibody
9. Positive screening test for rheumatoid factor
10. History of COVID-19
11. Positive FDA-authorized screening test for serum SARS-CoV-2 antibody or presence of SARS-CoV-2 on nasopharyngeal or oropharyngeal swab by FDA-authorized RT-PCR
12. History of allergy, anaphylaxis, or severe reaction to beef products (including milk and gelatin).

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2020-12-23 (Actual); Study Completion 2020-12-23 (Actual)

PRIMARY OUTCOMES:
Number of Participants Having Adverse Events | 29 Days
  Incidence and severity of other adverse events and severe adverse events (SAE)
Number of Participants Having Transfusion-Related Adverse Events | 29 Days
  transfusion-related adverse events

SECONDARY OUTCOMES:
Number of Participants Having Adverse Events | 90 Days
  Incidence and severity of adverse events and SAEs from Screening through Study Day 90
Pharmacokinetics from screening to day 90 | 90 Days
  SARS-CoV-2 binding (ELISA) and neutralizing (PRNT80) antibody titers from Screening through Study Day 90

CONTACTS AND LOCATIONS:
Overall Officials: David Hoover, MD, Principal Investigator — ICON GPHS
Locations (3):
- United States (3):
  - Alliance for Multispecialty Research, LLC, Wichita, Kansas
  - SUNY Upstate Medical University, Syracuse, New York
  - ICON Early Phase Services, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in the published article, after deidentification (test, tables, figures, and appendices)
Supporting Information: Study Protocol
Time Frame: Starting 6 months after publication and ending 36 months following article publication
Access Criteria: Anyone who wishes to access the data.